CLINICAL TRIAL: NCT04334915
Title: A Multicenter, Prospective, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of Cenicriviroc Mesylate on Arterial Inflammation in People Living With HIV
Brief Title: Study to Evaluate the Effects of Cenicriviroc Mesylate on Arterial Inflammation in People Living With HIV
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Industry supporter no longer supporting the study. Protocol A5415's study will run instead.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5363; 32389 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Cenicriviroc Mesylate (CVC) (Experimental): Cenicriviroc mesylate (CVC) 150 mg tablet once a day for at least 24 weeks will be added to the participants' pre-existing antiretroviral (ARV) regimens.
  For participants who are on an efavirenz (EFV)-based regimen, dosing will be 300 mg, administered as two 150-mg tablets, once a day.
  Interventions: Drug: Cenicriviroc Mesylate (CVC)
- Arm B: Placebo for CVC (Placebo Comparator): Placebo for CVC 150 mg tablet once a day for at least 24 weeks will be added to the participants' pre-existing ARV regimens.
  For participants who are on an EFV-based regimen, dosing will be 300 mg, administered as two 150-mg tablets, once a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenicriviroc Mesylate (CVC) — Administered orally
  Arms: Arm A: Cenicriviroc Mesylate (CVC)
Drug: Placebo — Administered orally
  Arms: Arm B: Placebo for CVC

SUMMARY:
The purpose of this study is to evaluate the effects of cenicriviroc mesylate (CVC) on arterial inflammation in people living with HIV.

DETAILED DESCRIPTION:
This study will evaluate the effects of cenicriviroc mesylate (CVC) on arterial inflammation in people living with HIV.

Participants will be randomized to either the CVC arm (Arm A) or placebo for CVC arm (Arm B). CVC 150 mg or placebo for CVC will be added to the participants' pre-existing antiretroviral (ARV) regimens once a day for at least 24 weeks. For participants who are on an efavirenz (EFV)-based regimen, dosing will be 300 mg once a day.

Study participants will remain on study treatment for approximately 24 weeks. Study visits may include blood collection, physical examinations, and FDG-PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load OR two HIV-1 RNA >1,000 copies/mL.

  * NOTE: The term "licensed" refers to a US Food and Drug Administration (FDA)-approved kit, which is required for all investigational new drug (IND) studies.
  * WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* Currently on a stable, continuous non-nucleoside reverse transcriptase inhibitor (NNRTI)-based or unboosted integrase strand transfer inhibitor (INSTI)-based antiretroviral therapy (ART) regimen for ≥48 weeks prior to study entry with no ART interruption longer than 7 consecutive days and with no plans to change ART during the course of the study.

  * NOTE A: Stable is defined as no within-class changes in ART regimen within 12 weeks prior to study entry and no between-class changes for 24 weeks prior to study entry.
  * NOTE B: Unboosted ART is defined as an ART regimen that does not include the pharmacologic booster COBI or RTV.
  * NOTE C: Modifications of ART formulation within 12 weeks prior to study entry (e.g., from standard formulation to fixed-dose combination of the same drugs), are permitted.
* Screening HIV-1 RNA level below the limit of quantification (e.g., <20, <40, <50, or <75 copies/mL, depending on the assay) using an FDA-approved assay with a quantification limit of 75 copies/mL or lower performed by any laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent within 90 days prior to study entry.
* All HIV-1 RNA levels within 48 weeks prior to study entry below the limit of quantification (e.g., <20, <40, <50, or <75 copies/mL, depending on the assay) using an FDA-approved assay with a quantification limit of 75 copies/mL or lower performed by any laboratory that has a CLIA certification or its equivalent.

  * NOTE A: Up to two HIV-1 RNA determinations that are between the assay quantification limit and 500 copies/mL (i.e., "blips") are allowed as long as the preceding and subsequent determinations are below the level of quantification.
  * NOTE B: The screening value may serve as the subsequent undetectable value following a blip.
* CD4+ cell count >200 cells/mm^3 obtained within 90 days prior to study entry at any US laboratory that has a CLIA certification or its equivalent.
* At least one of the following cardiovascular risk factors (current diagnosis or receiving treatment, except where a time period is specified):

  * Clinical atherosclerotic disease (symptomatic atherosclerotic lesions in any vessel)
  * Subclinical atherosclerotic disease (coronary artery calcification [CAC] >10 or presence of non-obstructive plaques)
  * DM or prediabetes (hemoglobin A1c [HbA1c] ≥5.7%) or impaired fasting glucose (documented fasting glucose of >100 mg/dL within 6 months prior to study entry) or insulin resistance (HOMA-IR ≥2.6) or any one of these laboratory values within 6 months prior to study entry
  * Obesity (body mass index [BMI] ≥30 kg/m^2) or enlarged iliac waist circumference (>40 inches in males, >35 inches in females)
  * NOTE: A BMI calculator is available at the Data Management Center (DMC) website: https://www.fstrf.org/ACTG/ccc.html
  * History of hypertension or blood pressure ≥130/80 mmHg measured during screening
  * NOTE: Blood pressure should be measured following the current ACTG Standardized Blood Pressure Measurement standard operating procedure (SOP). See the A5363 Manual of Procedures (MOPS) for the link to the SOP.
  * Elevated LDL cholesterol (fasting LDL of >160 mg/dL; result from sample taken within 90 days prior to study entry can be used)
  * Low HDL cholesterol (<40 mg/dL; result from sample taken within 90 days prior to study entry can be used)
  * Smoking (any current tobacco smoking)
  * Family history of premature CAD (first degree relative with CAD prior to age 55 for male relative and 65 for female relative; participant report is acceptable)
  * hsCRP >2.0 mg/L within 90 days prior to study entry without an active infection or acute illness at the time the sample was obtained
* The following laboratory values obtained within 90 days prior to study entry by any laboratory that has a CLIA certification or its equivalent.

  * Absolute neutrophil count (ANC) >750/mm^3
  * Platelet count >100,000/mm^3
  * Aspartate aminotransferase (AST) (SGOT) ≤5x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) (SGPT) ≤5x ULN
  * Alkaline phosphatase ≤5x ULN
  * Estimated glomerular filtration rate (GFR) ≥60 mL/min/1.73 m^2 as calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation
  * NOTE: See the A5363 MOPS for further information and a link to the CKD-Epi equation and calculator.
* Pre-entry FDG-PET/CT imaging (within 60 days prior to study entry) that has been deemed:

  * Interpretable as assessed by the central imaging core laboratory AND
  * Without incidental findings that will preclude participation in the study at the discretion of the site investigator
* For females of reproductive potential, negative serum or urine pregnancy test within 90 days prior to study entry and prior to starting study treatment at study entry by any clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care (POC)/CLIA-waived test.

  * NOTE: Reproductive potential is defined as girls who have reached menarche and women who have not been post-menopausal for at least 12 consecutive months with follicle-stimulating hormone (FSH) ≥40 IU/mL or 24 consecutive months if an FSH is not available, or have not undergone surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy).
* If participating in sexual activity that could lead to pregnancy, willingness of female participants to use two forms of contraception while receiving study medication and for 3 months after stopping study medication as required.

  * NOTE A: Acceptable forms of contraception include:
  * barrier methods (condoms [male or female] with or without a spermicidal agent, diaphragm, or cervical cap [with spermicide])
  * hormone-based contraception (oral, patch, parenteral, implants, or vaginal ring)
  * intrauterine device (IUD)
  * NOTE B: If the female participant is not of reproductive potential (women who are post-menopausal as defined above, or women who have undergone surgical sterilization [e.g., hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy]), she is eligible without requiring the use of a contraceptive method. Acceptable documentation of surgical sterilization and menopause is by participant-reported history.
* Men and women age ≥45 years.
* Ability and willingness of participant or legal guardian/representative to provide informed consent.

Exclusion Criteria:

* Acute coronary syndrome, defined as myocardial infarction (MI) or unstable angina, within 90 days prior to study entry.
* A current diagnosis of latent or active tuberculosis (TB) infection, any prior untreated TB infection, inadequate treatment of active TB, or inadequate treatment of latent TB.

  * NOTE A: Individuals with cases of active infection and latent TB infection with a history of adequate treatment may be considered for enrollment provided the individual has a negative chest X-ray following treatment and within 1 year prior to study entry.
  * NOTE B: Written documentation of prior TB treatment and negative chest x-ray is required.
* Current diagnosis with other intracellular pathogens (Mycobacterium avium complex, Listeria monocytogenes, Toxoplasma gondii, and Cryptococcus neoformans) within 90 days prior to study entry.
* Untreated hepatitis B virus (HBV) infection with detectable HBV DNA within 6 months prior to study entry.
* Current hepatitis C virus (HCV) infection (i.e., detectable HCV RNA within 6 months prior to study entry).
* Acute or clinically significant infection or illness requiring IV antibiotics or hospitalization within 90 days prior to study entry.
* History of cirrhosis with severe hepatic impairment and/or hepatic decompensation including ascites, hepatic encephalopathy, or variceal bleeding.
* Prior or planned liver transplantation.
* Active malignancy, except squamous cell skin cancer
* More than two HIV-1 RNA determinations ≥500 copies/mL within 48 weeks prior to study entry.
* Hemoglobin A1c >8% within 90 days prior to study entry by any laboratory that has a CLIA certification or its equivalent.
* Initiation of statin therapy or change in statin dose within 90 days prior to study entry.
* Current use of any of the statins at the doses indicated:

  * Atorvastatin, >20 mg/day dose
  * Lovastatin, >40 mg/day dose
  * Pitavastatin, >4 mg/day dose
  * Pravastatin, >40 mg/day dose
  * Rosuvastatin, ≥20 mg/day dose
  * Simvastatin, >40 mg/day dose
* Anticipated addition of any lipid lowering medication during the course of the study.
* Concurrent use of drugs with potential drug-drug interactions with CVC within 90 days prior to study entry (refer to the prohibited medications list in the study protocol).
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.
* Treatment within 30 days prior to study entry or anticipated treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons, cyclosporine, and tacrolimus).
* Immunization within 30 days prior to the pre-entry FDG-PET/CT imaging (refer to study protocol).
* History of radiation therapy.
* High radiation exposure within one year prior to entry, defined as having undergone more than two of any of the procedures below (includes having undergone the same procedure twice within one year prior to study entry):

  * Coronary artery catheterization with or without percutaneous coronary intervention (PCI)
  * Myocardial perfusion stress test
  * Coronary CT angiography
  * CT of the chest and abdomen
  * Barium enema
* Currently pregnant, breastfeeding, or planning to become pregnant during the length of the study and three months after completing the study.
* Body weight >300 pounds or >136 kilograms.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-22 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in arterial most diseased segment (MDS) 18F-fluorodeoxyglucose (FDG)-positron emission tomography (PET) target-to-background ratio (TBR), measured in the carotid arteries and aorta. | Pre-entry and week 24
  The standardized uptake value (SUV) of FDG will be measured in the carotid arteries, aortic root, and the left main coronary artery. The SUV is the decay-corrected tissue concentration of FDG (in kBq/mL) divided by the injected dose per body weight (kBq/g). TBR will be calculated for each vascular segment as the segment SUV divided by mean venous blood SUV. Change from baseline to week 24, where baseline is defined as pre-entry.

SECONDARY OUTCOMES:
Change in aortic TBR (and other TBRs) | Pre-entry and week 24
  Target-to-background ratio (TBR) will be calculated for each vascular segment as the segment standardized uptake value (SUV) divided by mean venous blood SUV. Change from baseline to week 24, where baseline is defined as pre-entry.
Change in SUV measured in the carotid arteries and aorta | Pre-entry and week 24
  The standardized uptake value (SUV) is the decay-corrected tissue concentration of fluorodeoxyglucose (FDG) (in kBq/mL) divided by the injected dose per body weight (kBq/g). Change from baseline to week 24, where baseline is defined as pre-entry.
Change in fasting glucose | Entry and week 24
  Change from baseline to week 24, where baseline is defined as entry.
Change in HOMA-IR | Entry and week 24
  Change from baseline to week 24, where baseline is defined as entry.
Change in sCD14 | Pre-entry, entry, week 22, and week 24
  Change from baseline to week 22/24, where baseline is defined as the average of pre-entry and entry values, and week 22/24 is defined as the average of week 22 and week 24 values.
Change in sCD163 | Pre-entry, entry, week 22, and week 24
  Change from baseline to week 22/24, where baseline is defined as the average of pre-entry and entry values, and week 22/24 is defined as the average of week 22 and week 24 values.
Change in IL-6 | Pre-entry, entry, week 22, and week 24
  Change from baseline to week 22/24, where baseline is defined as the average of pre-entry and entry values, and week 22/24 is defined as the average of week 22 and week 24 values.
Change in hsCRP | Pre-entry, entry, week 22, and week 24
  Change from baseline to week 22/24, where baseline is defined as the average of pre-entry and entry values, and week 22/24 is defined as the average of week 22 and week 24 values.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Lo, MD, MMSc, Study Chair — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https: https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.